CLINICAL TRIAL: NCT07313514
Title: The Value of the O-RADS Radiological Classification in Predicting the Malignancy of Ovarian Masses in Children
Acronym: MMO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9613
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ovarian; Mastopathy
Keywords: Malignancy in Ovarian Masses; Ovarian; Mastopathy
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When faced with an ovarian mass in a girl, conservative surgery (resection of the mass while preserving healthy ovarian tissue) via laparoscopy remains the most appropriate treatment option. However, this option is no longer indicated for malignant tumors, as this presents a risk of tumor dissemination that can significantly alter the child's subsequent prognosis. Therefore, for any malignant or suspected malignant tumor, radical treatment consisting of oophorectomy or salpingo-oophorectomy, often via laparotomy, is the standard. While keeping this therapeutic principle in mind, differentiating between benign and malignant entities remains the major challenge for clinicians. Furthermore, the diagnostic accuracy of the O-RADS classification based on MRI is not sufficiently established in the literature for children. Our project aims to conduct a multicenter study in the pediatric population to investigate the usefulness of this radiological classification in the preoperative diagnosis of ovarian masses.

ELIGIBILITY:
Inclusion Criteria:

* Girls under 16 years of age.
* Girls who underwent surgery for ovarian masses at the Pediatric Surgery Department of Mohammed VI University Hospital in Oujda during the study period.
* Girls who underwent surgery for ovarian masses at the Pediatric Surgery Department of Strasbourg University Hospital during the study period.
* Girls who underwent preoperative MRI.

Exclusion Criteria:

* Girls who underwent preoperative MRI.
* Patients who did not undergo surgery.
* Patients without histopathological examination of the surgical specimen.
* Patients without MRI as a preoperative diagnostic evaluation modality.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Girls under 16 years of age who underwent surgery for ovarian masses at the Pediatric Surgery Department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
O-RADS IRM (MRI) | Up to 9 months
  Score Interpretation Risk O-RADS MRI 1 Normal 0% O-RADS MRI 2 Benign < 1% O-RADS MRI 3 Probably Benign ~5% O-RADS MRI 4 Suspicious ~50% O-RADS MRI 5 Highly Suspicious > 90%

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Pédiatrique - CHU de Strasbourg - France, Strasbourg, France